CLINICAL TRIAL: NCT00780273
Title: Success Rate of Immediately Loaded Implants With Platform Switched Design Placed in the Anterior Part of the Mandible and Restored With Fixed Prostheses: a Randomized, Split-mouth, Masked, Prospective, Open, Comparison, Monocenter Trial
Brief Title: Success Rate of Immediately Loaded Implants With Platform Switched Design Placed in Anterior Part of Mandible and Restored With Fixed Prostheses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: DF 245
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Edentulism
Keywords: subjects with edentulous mandible

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ankylos dental implants. (Experimental): 3 Ankylos dental implants placed in platform switch configuration on one side of the mandible in support of a fixed restoration.
  A total number of 19 subjects participated in this randomized, split mouth, masked, prospective, open, comparison, monocenter study. Participants were subjects with an edentulous mandible who recieved 3 implants on each side which were splinted for the delivery of a fixed prosthesis.
  Interventions: Device: Ankylos Implants
- 3i Prevail dental implants. (Active Comparator): Three 3i Prevail dental implants placed on the opposite side of the mandible from the Ankylos implants in support of fixed dental restoration.
  After a baseline phase of 1 month the mandible sides of subjects were randomly assigned to one of the 2 parallel treatment groups: one side received ANKYLOS plus implants. The contralateral sde recieved Certain PREVAIL Implants. Abutments were installed and loaded immediately by a fixed temporary bridge. After 3 months the final prosthesis was incorporated.
  Interventions: Device: Biomet 3i Prevail Implants

INTERVENTIONS:
Device: Ankylos Implants — ANKYLOS Implant System vs Certain PREVAIL Implant
  Arms: Ankylos dental implants.
Device: Biomet 3i Prevail Implants
  Arms: 3i Prevail dental implants.

SUMMARY:
Change in crestal bone level implants at 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80
* male or female (female non-pregnant)
* sufficient oral hygiene
* no inflammation/disorder in the area of implant site
* edentulous mandible and sufficient prosthetic and conservative
* sufficient width and height of bone to place implants with diameters of 4.8mm and length of 11 mm
* provide written informed consent

Exclusion Criteria:

* demonstrate a need for pre-surgical bone or soft tissue augmentation in planned implant areas
* exhibit angulation requirements of restoration exceeding 15 degrees
* systemic metabolic disorder that would compromise post-operative tissue regeneration or osseointegration
* taking medication that would compromise post-operative healing and/or osseointegration
* bone disorders such as osteoporosis, hyperparathyroidism, Paget's disease, diabetes mellitus
* oncology treatment
* oral infection
* acute gingivitis and/or periodontitis
* local bone defects in the area of planned implantation
* disorders of oral mucosa (e.g., leukoplakia, oral lichen, pemphigoid lesions)
* received investigational drug within 30 days
* history of illicit drugs or alcohol abuse
* history of addiction to medication
* allergic to dental materials
* nicotine abuse (> 20 cigarettes/day)
* pregnant or nursing
* clinical significant or unstable medical or physiological conditions that would compromise participation in study
* unable or unwilling to return for follow-up visits for a period of 24 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Romanos, DDS, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Eastman Dept of Dentistry, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dental Implants.: 3 Ankylos dental implants placed in platform switch configuration on one side of the mandible in support of a fixed restoration.
  Ankylos Implants: ANKYLOS Implant System vs Certain PREVAIL Implant in split mouth study.
  A total of 19 subjects participated in this randomized, split-mouth, masked, prospective, open, comparison, monocenter study. Participants were subjects with an edentulous mandible who received 3 implants on each side which were splinted for the delivery of a fixed prosthesis.
  After a baseline phase of 1 month the mandible sides of subjects were randomly assigned to one of 2 parallel treatment groups: one side received ANKYLOS® plus Implants. The contralateral side received Certain® PREVAILTM Implants. Abutments were installed and loaded immediately by a fixed temporary bridge. After 3 months the final prosthesis was incorporated.
Period: Overall Study
Arm/Group | Dental Implants.
Started | 19
Completed | 17
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dental Implants.
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness - Treatment Difference in Mean Change in Crestal Bone Level
Description: Incidence of greater than 2 mm crestal bone (mesial or distal) loss. Reported in the percentage of analyzed implants.
Time Frame: 6 months after surgery
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Groups:
- Ankylos Dental Implants.: 3 Ankylos dental implants placed in platform switch configuration on one side of the mandible in support of a fixed restoration.
  Ankylos Implants: ANKYLOS Implant System vs Certain PREVAIL Implant
- 3i Prevail Dental Implants.: Three 3i Prevail dental implants placed on the opposite side of the mandible from the Ankylos implants in support of fixed dental restoration.
  Biomet 3i Prevail Implants
Arm/Group | Ankylos Dental Implants. | 3i Prevail Dental Implants.
Number analyzed (Participants) | 19 | 19
Number analyzed (Implants) | 52 | 53
Percentage of implants | 13 | 55

2. Primary Outcome: Effectiveness - Treatment Difference in Mean Change in Crestal Bone Level
Description: Incidence of greater than 2 mm crestal bone (mesial or distal) loss. Reported in the percentage of analyzed implants.
Time Frame: 12 months after surgery
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | Ankylos Dental Implants. | 3i Prevail Dental Implants.
Number analyzed (Participants) | 19 | 19
Number analyzed (Implants) | 49 | 50
Percentage of implants | 20 | 56

3. Primary Outcome: Effectiveness - Treatment Difference in Mean Change in Crestal Bone Level
Description: Incidence of greater than 2 mm crestal bone (mesial or distal) loss. Reported in the percentage of analyzed implants.
Time Frame: 24 months after surgery
Measure: Number; unit: Percentage of implants
Units Other Than Participants: Implants
Arm/Group | Ankylos Dental Implants. | 3i Prevail Dental Implants.
Number analyzed (Participants) | 19 | 19
Number analyzed (Implants) | 44 | 47
Percentage of implants | 11 | 70

ADVERSE EVENTS:
Groups:
- Dental Implants.: 3 Ankylos dental implants placed in platform switch configuration on one side of the mandible in support of a fixed restoration.
  Ankylos Implants: ANKYLOS Implant System vs Certain PREVAIL Implant in split mouth study.
Arm/Group | Dental Implants.
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No